CLINICAL TRIAL: NCT02553512
Title: Helius in Hypertension-I: The UK Hypertension Registry
Status: Completed | Type: Observational
Sponsor: Proteus Digital Health, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PB-HELIUS
Record Dates: First submitted 2015-09-15; First posted 2015-09-17 (Estimated); Results first posted 2017-06-16 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-04

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Ingestible Sensor and Wearable Sensor — This digital health offering passively acquires and records medication-taking and habits of daily living.

SUMMARY:
The purpose of this study is to demonstrate the use of a digital health offering in the management of persistent hypertension during chronic anti-hypertensive treatment.

DETAILED DESCRIPTION:
In patients with persistent essential systolic hypertension,who are undergoing assessment of their current pharmaceutical burden for blood pressure control, a digital health offering is used (1) to provide automatic and passive electronic documentation of medication adherence and patterns of medication taking, (2) to assist providers in distinguishing inadequate medication adherence or pharmacologic unresponsiveness as the root cause for persistent hypertension, and (3) to inform management decisions (dose adjustment, medication addition or substitution, adherence counseling, referral to a hypertension specialist).

Participating patients wear an adhesive Wearable Sensor ("Patch") continuously with replacement after one week, and ingest an inert tablet ("Pill") containing an Ingestible Sensor daily whenever they take their prescribed anti-hypertensive drugs.

The Patch automatically detects and records the dates and times of each "Pill" ingestion, daily step count, sleep duration and sleep interruptions, and the circadian pattern of rest and activity. After completion of each Patch's use, the recorded data are downloaded and incorporated into a report that includes blood pressures that are obtained at the time of clinic visits at the beginning and after 2 weeks of service use.

The final report is generated automatically and provided electronically to practitioners for review with their patient. The information that is obtained is incorporated by practitioners in advising next steps for blood pressure management.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of age ≥ 18 years
* Essential hypertension, consisting of:

  1. Blood pressure ≥150 or ≥90 during chronic treatment with 2 or more drugs for patients ≥80 years of age; or,
  2. Blood pressure ≥140 or≥90) during chronic treatment with 2 or more drugs for patients <80 years of age
* Ability to read and understand the instructions for participating
* Capacity to read and to speak English proficiently
* Capacity to provide informed consent

Exclusion Criteria:

* History of skin sensitivity to adhesive medical tape or metals
* History of acute or chronic dermatitis
* Any other condition that in the investigators opinion would compromise patient safety while participating
* Alcohol or other substance abuse
* Terminal illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having blood pressure (measured in mm Hg) ≥150 systolic or ≥90 diastolic during chronic treatment with 2 or more anti-hypertensive drugs, and age ≥80 years; or blood pressure ≥140 systolic or ≥90 diastolic during chronic treatment with 2 or more anti-hypertensive, and <80 years
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2013-09; Primary Completion 2014-12 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Godbehere, MD, Principal Investigator — North Brink Practice, Cambridgeshire UK

REFERENCES:
- [Background] Godbehere P, Wareing P. Hypertension assessment and management: role for digital medicine. J Clin Hypertens (Greenwich). 2014 Mar;16(3):235. doi: 10.1111/jch.12246. Epub 2014 Feb 5. No abstract available. PMID 24498940

RESULTS

PARTICIPANT FLOW:
Groups:
- Helius: Ingestible Sensor and Wearable Sensor
Period: Overall Study
Arm/Group | Helius
Started | 167
Completed | 144
Not Completed | 23

BASELINE CHARACTERISTICS:
Arm/Group | Helius
Number analyzed (Participants) | 151
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63
  Male | 88
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 151
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 151
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 151
Blood Pressure [Mean (Full Range); unit: mm Hg]
  Systolic | 154 [125 to 207]
  Diastolic | 88 [47 to 110]
Diabetes [Count of Participants; unit: Participants] | 45
Anti-Hypertensives (Type) [Count of Participants; unit: Participants]
  Generic | 136
  Generic and Branded | 15
  Branded | 0
Anti-Hypertensives (Number) [Count of Participants; unit: Participants]
  1 | 0
  2 | 93
  3-5 | 58
Anti-Hypertensives (Class) [Count of Participants; unit: Participants]
  ACE inhibitor | 82
  Angiotensin receptor blocker | 57
  Beta-blocker | 43
  Calcium channnel antagonist | 93
  Diuiretic | 72
  Fixed-dose combination | 3
  Other | 29

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Medication-taking (% Taking Adherence)
Description: Percent timing adherence is determined by the number of ingestion sensors detected by the wearable monitor, divided by the total number of ingestion sensors prescribed, for the 2 week-time frame.
Time Frame: 2 weeks
Measure: Median (Full Range); unit: percentage of taking adherence
Arm/Group | Helius
Number analyzed (Participants) | 151
percentage of taking adherence | 75 [53 to 100]

2. Primary Outcome: Pattern of Medication-taking (% Scheduling Adherence)
Description: Percent scheduling adherence is determined by the number of ingestion sensors detected within a ± 2-hour time window around the prescribed dosing period, divided by the number of ingestion sensors detected by the wearable sensor during that dosing period, over the 2-week time frame.
Time Frame: 2 weeks
Measure: Median (Full Range); unit: percentage of scheduling adherence
Arm/Group | Helius
Number analyzed (Participants) | 151
percentage of scheduling adherence | 65 [21 to 100]

3. Secondary Outcome: Proportion of Patients Capable of Achieving Blood Pressure Control on Existing Treatment
Description: Percentage of participants
Time Frame: 2 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Helius
Number analyzed (Participants) | 151
percentage of participants | 32

4. Secondary Outcome: Change in Systolic and Diastolic Blood Pressure After Use of Digital Health Offering
Description: Decrease in systolic and diastolic blood pressure (measured in mm Hg) after 2 weeks when compared to baseline
Time Frame: 2 weeks
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Helius
Number analyzed (Participants) | 151
mm Hg
  Systolic | 9.7 [7.0 to 12.5]
  Diastolic | 5.0 [3.5 to 6.5]

5. Secondary Outcome: Blood Pressure Management After Use of Digital Health Offering
Description: Summary of provider actions following review of final report with patient (dose or medication change, adherence counseling, referral to a hypertension specialist)
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Helius
Number analyzed (Participants) | 151
Participants
  Meds review/Adherence counseling/no med changes | 122
  Antihypertensive medication change | 19
  No further action taken | 10

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Helius
All-Cause Mortality (participants affected / at risk) | 0/151
Serious Adverse Events (participants affected / at risk) | 0/151
Other Adverse Events (participants affected / at risk) | 18/151
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Helius (N=151)
Rash (Skin and subcutaneous tissue disorders) | 12
Gastrointestinal complaint (Gastrointestinal disorders) | 6

LIMITATIONS AND CAVEATS:
This was an open-label registry. Patients may have increased their adherence due to a Hawthorne effect. Patients may have been selective in the medications that they actually ingested.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No